CLINICAL TRIAL: NCT05839678
Title: How to Differentiate and Treat Cystic Laesions in the Anterior Mediastinum (DETECTION)
Acronym: DETECTION
Status: Recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Erasmus Medical Center (Other); The Netherlands Cancer Institute (Other)
Responsible Party: Principal Investigator, Florit Marcuse, Principal investigator, MD PhD, Maastricht University Medical Center
Other Study IDs: 2022-3413
Record Dates: First submitted 2023-04-20; First posted 2023-05-03 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Cysts
MeSH Terms: conditions — Cysts

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multicenter trial about anterior mediastinal cysts

ELIGIBILITY:
Inclusion Criteria: cysts in the anterior mediastinum

* Thymic cysts
* Bronchogenic cysts
* Pericardial cysts
* Cystic thymoma
* Cystic teratoma

Exclusion Criteria:

* Patients <18 years old
* Patients without radiological imaging
* Patients without approval for follow-up

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with cysts in the anterior mediastinum
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Percentage correctly diagnosed cystic laesions | 2000-2022

SECONDARY OUTCOMES:
Patient characteristics, complications, comborbidities | 2000-2022

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht UMC, Maastricht, Limburg, Netherlands